CLINICAL TRIAL: NCT05634187
Title: Simultaneous Evaluation of Endoscopic Features in Patients Suffering From Gastroesophageal Reflux: Functional Endoscopy Gives Insight for ENT (Ear-nose-throat) and GI Alterations - a Prospective Study
Brief Title: One-stop-shop Endoscopy in Reflux-patients: Evaluation of ENT and GI Features
Acronym: ENTGI-reflux
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: Endoscopy_ENT-GI-Reflux
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-01

CONDITIONS: Reflux Disease; Reflux, Gastroesophageal; Reflux, Laryngopharyngeal
Keywords: functional endoscopy
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngopharyngeal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering from symptoms suggestive for gastroesophageal reflux disease: Patients suffering from dysphasia, heartburn, laryngitis or pharyngitis suggestive for gastroesophageal reflux disease
  Interventions: Device: Functional endoscopy

INTERVENTIONS:
Device: Functional endoscopy — Transnasal endoscopy by an ultrathin video endoscope

SUMMARY:
Patients suffering from gastroesophageal reflux may suffer from both esophageal and laryngeal irritations. The investigators developed an endoscopic technique called functional endoscopy to evaluate alterations in the larynx and pharynx as well as in the esophagus simultaneously as one-stop-shop.

DETAILED DESCRIPTION:
Patients suffering from gastroesophageal reflux may present to a variety of medical specialists according to their individual complaints (e.g., heartburn, hoarseness, dysphasia). In general, these addressed specialist may focus their attention to their individual fields of interest.

The investigators developed an endoscopic technique called functional endoscopy to evaluate patients with various GI- or ENT (ear-nose-throat)-symptoms being suggestive for gastroesophageal reflux disease.

In functional endoscopy, unsedated patients are examined with an ultrathin endoscope via the transnasal route. Reflux-associated features in the field of interest of the ENT-doctor and the GI-specialist are recorded and documented in the same session.

ELIGIBILITY:
Inclusion Criteria:

- Patients suffering from dysphasia, heartburn, laryngitis or pharyngitis suggestive for gastroesophageal reflux disease

Exclusion Criteria:

* Age under 18 years
* Inability to understand information for participation
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from dysphasia, heartburn, laryngitis or pharyngitis suggestive for gastroesophageal reflux disease
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Endoscopic findings in the laryngeal and pharyngeal area due to reflux | 30 minutes
  Assessment of endoscopic findings in the laryngeal and pharyngeal area
Endoscopic findings in the oesophagus due to reflux | 30 minutes
  Assessment of endoscopic findings in the oesophagus

SECONDARY OUTCOMES:
Safety of procedure | 30 minutes
  Assessments of complications

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Domagk, MD, Study Chair — Josephs Hospital Warendorf, Academic Teaching Hospital University of Muenster
Locations (1):
- University of Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheung J, Bailey R, Veldhuyzen van Zanten S, McLean R, Fedorak RN, Morse J, Millan M, Guzowski T, Goodman KJ; CANHelp working group. Early experience with unsedated ultrathin 4.9 mm transnasal gastroscopy: a pilot study. Can J Gastroenterol. 2008 Nov;22(11):917-22. doi: 10.1155/2008/323027. PMID 19018337
- [Result] Herrmann IF, Scarpignato C. [Functional endoscopy : the physiological and pathophysiological basis of reflux disease, diagnosis and therapy]. HNO. 2009 Dec;57(12):1221-36. doi: 10.1007/s00106-009-1934-z. German. PMID 19924362
- [Result] Herrmann IF, Gadebusch Bondio M, Domagk D, Strahl M, Arens C. [New possibilities with retroflexed functional endoscopy]. HNO. 2018 Jul;66(7):527-533. doi: 10.1007/s00106-018-0518-1. German. PMID 29968191
- [Result] Ruckert J, Lenz P, Heinzow H, Wessling J, Warnecke T, Herrmann IF, Strahl M, Lenze F, Nowacki T, Domagk D. Functional endoscopy in neurogenic dysphagia: a feasibility study focusing on the esophageal phase of swallowing. Endosc Int Open. 2021 Apr;9(4):E646-E652. doi: 10.1055/a-1380-3224. Epub 2021 Apr 15. PMID 33880400